CLINICAL TRIAL: NCT01580969
Title: A Phase 1b/2 Study of Repeat rAdiation, Minocycline, and Bevacizumab in Patients With Recurrent gliOma (RAMBO)
Brief Title: Repeat Radiation, Minocycline and Bevacizumab in Patients With Recurrent Glioma
Acronym: RAMBO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCI55264
Record Dates: First submitted 2012-03-06; First posted 2012-04-19 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Glioma
Keywords: glioma
MeSH Terms: conditions — Glioma | interventions — Bevacizumab; Minocycline; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 0: 100 mg bid (Experimental): Patients receiving minocycline 100 mg bid, bevacizumab, and radiation therapy.
  Interventions: Drug: Bevacizumab; Drug: Minocycline; Radiation: Radiation
- Dose Level 1: 200 mg bid (Experimental): Patients receiving minocycline 200 mg bid, bevacizumab, and radiation therapy.
  Interventions: Drug: Bevacizumab; Drug: Minocycline; Radiation: Radiation
- Dose Level 2: 400 mg bid (Experimental): Patients receiving minocycline 400 mg bid, bevacizumab, and radiation therapy.
  Interventions: Drug: Bevacizumab; Drug: Minocycline; Radiation: Radiation

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered in accordance with the FDA-approved dose for gliomas, 10mg/kg IV every 2 weeks. Bevacizumab will be continued every two weeks as long as tolerated. One cycle of bevacizumab will be 28 days, with treatments on day1 and day 15.
  Other Names: Avastin
Drug: Minocycline — Minocycline will be given by mouth twice a day at the assigned dose level. Minocycline will be started on the day prior to radiation and continued until progression or intolerance.
Radiation: Radiation — Radiation planning will be individualized by the radiation oncologist based on the location of the current radiation field relative to prior radiation doses. The length and fractionation will be determined individually by the radiation oncologist.

SUMMARY:
The primary objective of step 1 is the rate of adverse events of minocycline and bevacizumab during reirradiation and of step 2 is the response rate to bevacizumab, reirradiation, and minocycline. The secondary objectives are the response rate, Progression Free Survival (PFS)-3, PFS-6, and effects on quality of life and cognition from repeat radiation and bevacizumab.

DETAILED DESCRIPTION:
After providing informed consent, patients will undergo screening for eligibility to participate in the study. Screening will start within 21 days prior to dosing.

Subjects will have an MRI within 21 days of starting radiation. QOL and cognition measures will be performed within 21 days of starting radiation. Radiation will be given with parameters determined on an individual basis by the radiation oncologist. Bevacizumab will be continued at 10mg/kg IV every 2 weeks. Minocycline will be given twice a day starting at 100mg PO bid. MRI, QOL, and cognitive tests will be obtained 1, 3 and 6 months after the end of radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old with a life expectancy of at least 8 weeks
2. Radiographically proven recurrent (≥ first relapse), intracranial glioma
3. Previous treatment with external beam radiation
4. Radiographic progression on current or prior bevacizumab treatment
5. Women of child-bearing potential must have a negative pregnancy test within 7 days of initiation of dosing and must agree to use an acceptable method of birth control while on study drug and for 3 months after the last dose. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year. Men of child-bearing potential must also agree to use an acceptable method of birth control while on study drug, and for 3 months after the last dose.
6. Karnofsky performance status of ≥50
7. Adequate hematologic, hepatic, and renal function (absolute neutrophil count ≥1.0 x 109/L, Hgb >9 g/dL, platelet count ≥50 x 109/L, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5x ULN, creatinine ≤1.5x ULN)
8. Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements
9. Systolic blood pressure ≤ 160 mg Hg or diastolic pressure ≤ 90 mg Hg within 14 days prior to study registration
10. Prothrombin time/international normalized ratio (PT INR) < 1.4 for patients not on warfarin confirmed by testing within 14 days prior to study registration
11. Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight (LMW) heparin) must have no active bleeding or pathological condition that carries a high risk of bleeding, and must be on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin

Exclusion Criteria:

1. Use of an investigational drug within 14 days or within 5 half-lives of teh investigational drug, whichever is shorter
2. Progression within 3 months of previous radiation by Radiographic Assessment in Neurooncology (RANO) criteria
3. History of Grade 2 (CTCAE v4) or greater acute intracranial hemorrhage
4. A concurrent active cancer that requires non-surgical therapy (e.g. chemotherapy, radiation, adjuvant therapy).
5. Patients with serious illnesses, uncontrolled infection, medical conditions, or other medical history including abnormal laboratory results, which in the investigator's opinion would be likely to interfere with a patient's participation in the study, or with the interpretation of the results
6. Women of child-bearing potential who are pregnant or breast feeding
7. Unstable angina and/or congestive heart failure in the last 6 months, transmural myocardial infarction within the last 6 months, New York Heart Association grade II or higher congestive heart failure requiring hospitalization within 12 months prior to registration, evidence of recent myocardial infarction by EKG performed within 14 days of registration, serious or inadequately controlled cardiac arrhythmia, significant vascular and peripheral vascular disease, evidence of bleeding diathesis or coagulopathy
8. History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months
9. Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for tumor resection
10. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
11. Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07-06 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cohen, MD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Started | 6 | 3 | 13
Completed | 3 | 3 | 13
Not Completed | 3 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid | Total
Number analyzed (Participants) | 6 | 3 | 13 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 11 | 18
  >=65 years | 1 | 1 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.33 (14.45) | 61 (11.27) | 51.69 (16.13) | 53.95 (14.87)
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 74] | 55 [54 to 74] | 53 [31 to 76] | 55.5 [31 to 76]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 2 | 3 | 9 | 14
  Female | 3 | 0 | 4 | 7
  Not Reported | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 2 | 12 | 19
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 2 | 13 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse Events were assessed from start of minocycline treatment (one day prior to start of radiation therapy) until 28 days following the end of radiation therapy. Adverse events were assessed using the Common Terminology for Adverse Events (CTCAE) version 4.0. Each event was assigned a grade (1-5), with lower grades indicating milder events. Events were categorized as severe (grade 3-4) or non-severe (grade 1-2). All adverse events were recorded, regardless of attribution to study treatment. Reported below are the number of patients who experienced any non-severe AE and the number of patients who experienced any severe AE. A full listing of AEs (severe and non-severe) are listed in the Adverse Events module of the Results section.
Time Frame: From first dose of study treatment to 28 days following radiation therapy (7-8 weeks)
Population: In dose level 0, three patients were withdrawn prior to completing the reporting period for the primary objective, making them unevaluable, and they were replaced.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 3 | 3 | 13
Participants
  Any Severe (G3-4) Adverse Event | 0 | 1 | 3
  Any Non-Severe (G1-2) Adverse Event | 3 | 3 | 11

2. Secondary Outcome: Progression Free Survival (PFS) at 3 Months
Description: Proportion of patients who have not progressed 12 weeks after the end of radiation therapy. Radiographic Assessment in Neurooncology (RANO) criteria will be used to assess progression and response. Estimates were done by Kaplan-Meier methods to account for patients whose data was censored prior to progression.
Time Frame: From start of study treatment until 12 weeks after radiation therapy (15-16 weeks)
Population: Patients who did not complete the Dose Limiting Toxicity (DLT) evaluation period (3 patients in Dose Level 0) were excluded from PFS analysis.
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 3 | 3 | 13
probability of survival | 1.000 [1.00 to 1.00] | 0.667 [0.2995 to 1.00] | 0.646 [0.418 to 0.998]

3. Secondary Outcome: Progression Free Survival (PFS) at 6 Months
Description: Proportion of patients who have not progressed 26 weeks after the end of radiation therapy. Radiographic Assessment in Neurooncology (RANO) criteria will be used to assess progression and response. Estimates were done by Kaplan-Meier methods to account for patients whose data was censored prior to progression.
Time Frame: From start of study treatment until 26 weeks after radiation therapy (29-30 weeks)
Population: Patients who did not complete the DLT period (3 patients in Dose Level 0) were excluded from PFS analysis.
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 3 | 3 | 13
probability of survival | 0.667 [0.2995 to 1.00] | 0.333 [0.0673 to 1.00] | 0.277 [0.106 to 0.723]

4. Secondary Outcome: Tabulation of Tumor Best Responses
Description: Tabulation of the best tumor response participants achieved from baseline through 26 weeks after the end of radiation therapy. Radiographic Assessment in Neurooncology (RANO) criteria will be used to assess progression and response.
Time Frame: From start of study treatment until 26 weeks after radiation therapy (29-30 weeks)
Population: In Dose Level 0, three patients did not complete any follow-up scans and were excluded from analysis. In Dose Level 2, six patients did not complete any follow-up scans and were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 3 | 3 | 7
Participants
  Complete Response | 1 | 0 | 0
  Partial Response | 0 | 1 | 0
  Stable Disease | 2 | 1 | 5
  Progressive Disease | 0 | 1 | 1
  Not Evaluable per RANO Criteria | 0 | 0 | 1

5. Secondary Outcome: Quality of Life Change Over Time
Description: The M. D. Anderson Symptom Inventory - Brain Tumors (MDASI-BT) scale was used to assess patients at baseline, 4 weeks post-radiation, 12 weeks post-radiation, and 26 weeks post-radiation. Means and standard deviations from baseline and 26 post-radiation are reported here. MDASI-BT is a 28 item assessment using a 0-10 scale. Part 1 contains 22 items and assesses severity of symptoms, with a score range from 0 to 220. Part 2 contains 6 items and assesses the degree to which symptoms interfere with daily life, with a score range from 0 to 60. The Total score adds Part 1 and Part 2 together to assess total symptom burden, with a score range from 0 to 280. For all parts of the assessment, higher scores indicate a lower quality of life and worse symptom burden.
Time Frame: From start of study treatment until 26 weeks after radiation therapy (29-30 weeks)
Population: 22 patient completed the baseline questionnaire, and 4 patients completed the 26 week post-radiation questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 6 | 3 | 13
units on a scale
  Baseline - Part 1 Score | 45.83 (33.43) | 29.67 (18.77) | 39.08 (24.23)
  Baseline - Part 2 Score | 15.67 (12.61) | 11.67 (7.51) | 16.85 (15.38)
  Baseline - Total Score | 61.5 (43.91) | 41.33 (24.09) | 55.92 (37.78)
  26 Week Post Radiation - Part 1 Score: number analyzed (Participants) | 2 | 1 | 1
  26 Week Post Radiation - Part 1 Score | 48 (0) | 55 (NA) — Standard deviation not calculated for single participant | 14 (NA) — Standard deviation not calculated for single participant
  26 Week Post Radiation - Part 2 Score: number analyzed (Participants) | 2 | 1 | 1
  26 Week Post Radiation - Part 2 Score | 22 (12.73) | 29 (NA) — Standard deviation not calculated for single participant | 15 (NA) — Standard deviation not calculated for single participant
  26 Week Post Radiation - Total Score: number analyzed (Participants) | 2 | 1 | 1
  26 Week Post Radiation - Total Score | 70 (12.73) | 84 (NA) — Standard deviation not calculated for single participant | 29 (NA) — Standard deviation not calculated for single participant

6. Secondary Outcome: Cognitive Change Over Time - DET
Description: The Cogstate software was used to assess cognitive function at baseline, 4 weeks post-radiation, 12 weeks post-radiation, and 26 weeks post-radiation. Mean scores and standard deviations from baseline and 26 weeks post-radiation are reported here. Detection Test (DET) measures sensory registration, vigilance, and reaction time. DET is scored based on the speed of performance: mean of the log10 transformed reaction time for correct responses [measured in log10 milliseconds (MS)]. Lower scores meant a better performance.
Time Frame: From start of study treatment until 26 weeks after radiation therapy (29-30 weeks)
Population: 14 patients completed the baseline assessment and 3 patients completed the 26 weeks post radiation therapy assessment. Patients were not required to complete the Cogstate assessment if they took more than one hour to complete it, or if they could not operate a computer or if they could not complete the practice tests.
Measure: Mean (Standard Deviation); unit: log10 ms
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 5 | 3 | 6
log10 ms
  Baseline | 2.72 (0.2) | 2.51 (.1) | 2.62 (0.11)
  26 Weeks Post Radiation: number analyzed (Participants) | 1 | 1 | 1
  26 Weeks Post Radiation | 2.79 (NA) — Standard deviation not calculated for single participant | 2.9 (NA) — Standard deviation not calculated for single participant | 2.67 (NA) — Standard deviation not calculated for single participant

7. Secondary Outcome: Cognitive Change Over Time - IDN
Description: The Cogstate software was used to assess cognitive function at baseline, 4 weeks post-radiation, 12 weeks post-radiation, and 26 weeks post-radiation. Mean scores and standard deviations from baseline and 26 weeks post-radiation are reported here. Identification Test (IDN) measures basic information processing and decision speed. IDN is scored based on the speed of performance: mean of the log10 transformed reaction time for correct responses [measured in log10 milliseconds (MS)]. Lower scores meant a better performance.
Time Frame: From start of study treatment until 26 weeks after radiation therapy (29-30 weeks)
Population: 16 patients completed the baseline assessment and 3 patients completed the 26 weeks post radiation therapy assessment. Patients were not required to complete the Cogstate assessment if they took more than one hour to complete it, or if they could not operate a computer or if they could not complete the practice tests.
Measure: Mean (Standard Deviation); unit: log10 MS
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 5 | 3 | 8
log10 MS
  Baseline | 2.86 (0.08) | 2.72 (0.05) | 2.78 (0.07)
  26 Weeks Post Radiation: number analyzed (Participants) | 1 | 1 | 1
  26 Weeks Post Radiation | 2.89 (NA) — Standard deviation not calculated for single participant | 2.97 (NA) — Standard deviation not calculated for single participant | 2.78 (NA) — Standard deviation not calculated for single participant

8. Secondary Outcome: Cognitive Change Over Time - OCLT
Description: The Cogstate software was used to assess cognitive function at baseline, 4 weeks post-radiation, 12 weeks post-radiation, and 26 weeks post-radiation. Mean scores and standard deviations from baseline and 26 weeks post-radiation are reported here. One Card Learning Test (OCLT) measures visuoperceptual learning and memory. OCLT is a score defined as the arcsine transformation of the square root of the proportion of correct responses to 80 OCLT questions. The transformed score ranges from 0 to 1.5708 where a higher score means better performance.
Time Frame: From start of study treatment until 26 weeks after radiation therapy (29-30 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Arcsine [(sqrt) proportion correct]
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 5 | 3 | 8
Arcsine [(sqrt) proportion correct]
  Baseline | 0.95 (0.18) | 0.91 (0.23) | 0.85 (0.15)
  26 Weeks Post Radiation: number analyzed (Participants) | 1 | 1 | 1
  26 Weeks Post Radiation | 0.94 (NA) — Standard deviation not calculated for single participant | 0.71 (NA) — Standard deviation not calculated for single participant | 0.96 (NA) — Standard deviation not calculated for single participant

9. Secondary Outcome: Cognitive Change Over Time - GMLT
Description: The Cogstate software was used to assess cognitive function at baseline, 4 weeks post-radiation, 12 weeks post-radiation, and 26 weeks post-radiation. Mean scores and standard deviations from baseline and 26 weeks post-radiation are reported here. Groton Maze Learning Test (GMLT) measures special learning and executive functioning, including working memory, error monitoring, and ability to integrate feedback to modify problem solving. GMLT score is the number of errors made (lower score indicates better performance).
Time Frame: From start of study treatment until 26 weeks after radiation therapy (29-30 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
Number analyzed (Participants) | 5 | 3 | 8
errors
  Baseline | 96.4 (31.17) | 90.67 (38.55) | 84.38 (31.46)
  26 Weeks Post Radiation: number analyzed (Participants) | 1 | 1 | 1
  26 Weeks Post Radiation | 61 (NA) — Standard deviation not calculated for single participant | 87 (NA) — Standard deviation not calculated for single participant | 48 (NA) — Standard deviation not calculated for single participant

ADVERSE EVENTS:
Time Frame: AEs were collected starting with the first dose of minocycline treatment until the last dose of study treatment. Serious Adverse Events (SAEs) continued to be collected until 30 days after last dose of study treatment.
Description: The occurrence of adverse events was sought by non-directive questioning of the patient at each visit or phone contact during the study. Adverse events also may have been detected when they were volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Dose Level 0: 100 mg Bid | Dose Level 1: 200 mg Bid | Dose Level 2: 400 mg Bid
All-Cause Mortality (participants affected / at risk) | 2/6 | 0/3 | 2/13
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/3 | 8/13
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0: 100 mg Bid (N=6) | Dose Level 1: 200 mg Bid (N=3) | Dose Level 2: 400 mg Bid (N=13)
Confusion (Psychiatric disorders) | 0 | 0 | 1
Death NOS (General disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 3 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0: 100 mg Bid (N=6) | Dose Level 1: 200 mg Bid (N=3) | Dose Level 2: 400 mg Bid (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 (4)
Ataxia (Nervous system disorders) | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 2
Concentration impairment (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 (5)
Cushingoid (Endocrine disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 (2) | 5
Depression (Psychiatric disorders) | 0 | 0 | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 5 (6)
Dizziness (Nervous system disorders) | 1 | 1 | 8 (13)
Dysarthria (Nervous system disorders) | 0 | 1 | 2 (3)
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (4)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 4
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eye disorders - Other (Eye disorders) | 2 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 3
Fatigue (General disorders) | 3 (5) | 1 | 5 (8)
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 2 | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 1
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 (5) | 2
Hemoglobin increased (Investigations) | 1 (2) | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 (3) | 2 (7) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 2 (6)
Irritability (General disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 4
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 7 (12)
Nervous system disorders - Other (Nervous system disorders) | 0 | 1 (2) | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (2)
Rhinitis infective (Infections and infestations) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 (3) | 5 (9)
Weight gain (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 1 | 1 (3) | 2 (3)
White blood cell decreased (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT01580969/Prot_SAP_000.pdf